CLINICAL TRIAL: NCT06026969
Title: Pregnancy and Early Neurodevelopmental Outcomes Following In Utero Lyme Disease Exposure
Status: Recruiting | Type: Observational
Sponsor: Children's National Research Institute (Other)
Collaborators: Clinical Trials Network for Lyme and Other Tick-Borne Diseases (Unknown); Steven & Alexandra Cohen Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 00000425
Record Dates: First submitted 2023-08-15; First posted 2023-09-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Lyme Disease; Post-Treatment Lyme Disease; Chronic Lyme Disease; Tick-Borne Infections; Pregnancy Complications; Child Development
MeSH Terms: conditions — Lyme Disease; Post-Lyme Disease Syndrome; Tick-Borne Diseases; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lyme disease: Pregnant participants in the "Lyme disease" cohort will meet CDC criteria for clinical and/or laboratory diagnosis of Lyme disease during pregnancy based on stage of disease. Participants will be enrolled following confirmation that they have been diagnosed by a medical professional per CDC guidelines.
  Participants in this cohort may be enrolled during any trimester of pregnancy. Live-born infants will be included in the cohort and followed through age 18 months.
  Interventions: Other: Neurodevelopmental assessments and follow-up
- Post-treatment Lyme Disease Syndrome (PTLDS) or Chronic Lyme: Pregnant participants in the "PTLDS/Chronic Lyme" cohort will have been diagnosed with PTLDS/Chronic Lyme by a health care provider no less than 6 months, but no greater than 3 years, prior to enrollment. Participants will be enrolled following confirmation that they have been diagnosed by a medical professional per CDC guidelines.
  Participants in this cohort may be enrolled during any trimester of pregnancy. Live-born infants will be included in the cohort and followed through age 18 months.
  Interventions: Other: Neurodevelopmental assessments and follow-up

INTERVENTIONS:
Other: Neurodevelopmental assessments and follow-up — All infants included in this study will receive standardized neurodevelopmental assessment and neurological examinations through age 18 months.

SUMMARY:
The purpose of this pilot study is to assess the feasibility of longitudinal neurodevelopmental evaluation of fetuses and infants exposed to Lyme disease in utero. Participants with Lyme disease or Post-Treatment Lyme Disease Syndrome (PTLDS) will be recruited during pregnancy. Pregnancies will be monitored and infant development will be assessed from birth until age 18 months.

DETAILED DESCRIPTION:
Childhood neurodevelopmental outcomes following antenatal Lyme disease exposure are not yet known. This pilot study will lay the groundwork for a larger study to determine the effect of in utero exposure to Lyme disease on pregnancy and early childhood neurodevelopmental outcomes. Understanding the effects on the developing brain is essential in order to inform timely prenatal and postnatal treatments to protect the fetus exposed to Lyme disease during pregnancy. Once childhood neurodevelopmental outcomes are known, appropriate follow-up and treatment guidelines can be developed to help better support children's developmental needs.

The primary aim of this study is to assess the feasibility of longitudinal follow-up of fetuses and infants exposed to Lyme disease in utero.Lyme disease in pregnancy and the impact on the fetus/child following in utero exposure has been identified as a priority research area; this pilot study is the essential step to plan a large study that will fill this knowledge gap and make a substantial contribution to the field.

The investigators will perform a prospective pilot longitudinal cohort study of B. burgdorferi-infected parents and their in-utero-exposed fetuses/infants. Patients included in this study will have a clinical diagnosis of Lyme disease during gestation or have been diagnosed with Lyme disease and/or PTLDS within 3 years preceding pregnancy.

Pregnant participants will receive a fetal MRI and ultrasound during the second or third trimesters of gestation. The investigators will conduct optional qualitative interviews with interested participants during their 3rd trimester to gather additional data on their experiences with Lyme disease/PTLDS during pregnancy. The placenta will be collected at birth and analyzed by an experienced placental pathologist per a standard protocol. Parent and infant blood will be tested for Lyme disease serology and markers of inflammation.

Following birth, infants will receive an unsedated brain MRI and a cranial ultrasound. The investigators will complete serial developmental evaluations using standardized assessments at multiple timepoints through age 18 months and receive neurological examinations. Throughout the study, participants will also be asked to complete questionnaires including but not limited to topics such as medical history, nutrition, breastfeeding, and socioeconomic information.

ELIGIBILITY:
Inclusion Criteria:

* English speaker
* Currently reside in the United States or Canada
* Meet CDC criteria for: (1) clinical and/or laboratory diagnosis of Lyme disease during any stage of current pregnancy, OR (2) clinical diagnosis of PTLDS/Chronic Lyme within 3 years of current pregnancy
* Able to be contacted for follow-up

Exclusion Criteria:

* Intellectually unable to comprehend study procedures
* Health issues or metallic implant that precludes undergoing MRI
* Incapable of completing study requirements (note: inability to travel to Children's National for in-person follow-up [for example, due to bedrest, travel restrictions, or financial inability to travel] is NOT an exclusion criterion; any interested and eligible participants requiring "remote only" participation will be permitted to join the study and complete all requirements besides in-person follow-up)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant participants with confirmed Borrelia burgdorferi infection or diagnosed PTLDS/Chronic Lyme will be enrolled during any trimester of pregnancy. All live-born infants will be followed to age 18 months and included in the study regardless of birth outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of parent-infant dyads enrolled in the study through completion of their infant's 18-month follow-up visit | 7/1/2023 - 6/30/2025
  The primary outcome of this pilot study is to assess the feasibility of enrollment and longitudinal follow-up of Lyme-exposed dyads. Investigators will measure the number of parent-infant dyads who are eligible for participation, who participate in each study visit, and who successfully complete the study through infant age 18 months, throughout the duration of the study.

SECONDARY OUTCOMES:
Warner Initial Developmental Evaluation (WIDEA) | Child ages: 2 months, 6 months, 12 months, 18 months
  Infants will be evaluated at 2, 6, 12, and 18 months of age using the Warner Initial Developmental Evaluation (WIDEA). The WIDEA is a 43-item questionnaire to assess the functional domains of self-care, motor function, communication, and social cognition in young children.
Ages and Stages Questionnaire (ASQ) | Child ages: 2 months, 6 months, 12 months, 18 months
  Infants will be evaluated at 2, 6, 12, and 18 months of age using the Ages and Stages Questionnaire (ASQ). The ASQ will assess for possible developmental delays in the domains of communication, gross motor, fine motor, problem solving, and personal adaptive skills.
Alberta Infant Motor Scale (AIMS) | Child ages: 2 months, 6 months, 12 months, 18 months
  Infants will be evaluated at 2, 6, 12, and 18 months of age using the Alberta Infant Motor Scale (AIMS). The AIMS is an observational motor assessment that can be done in-person or using telehealth.
Infant height | All study visits between birth - 18 months of age
  Infants' height in centimeters will be collected at each study visit.
Infant weight | All study visits between birth - 18 months of age
  Infants' height in kilograms will be collected at each study visit.
Infant head circumference | Birth - 18 months of age
  Infants' head circumference in centimeters will be collected at each study visit.
Placental tissue analysis | Placenta to be collected at delivery hospital immediately after birth
  The placenta will be collected at birth and analyzed by an experienced placental pathologist per a standard protocol. The study team will provide the pregnant participant a letter about their study participation that they can share with their obstetrician requesting placental pathology to be performed. The study coordinator will request the paraffin embedded blocks and/or slides to be sent to Children's National for additional analysis including silver stain. Silver stain will be included to identify any spirochetes in placental tissue.
Analysis of parent and infant blood | Adult: during pregnancy between 20-38 weeks gestational age, and between infant age 2-8 weeks; Child: Between ages 2-8 weeks
  Blood will be collected at the study visit in the Lyme-exposed parent and infant to measure Lyme serology (IgM, IgG), PCR, and inflammatory cytokines. The pregnant participant will have two blood draws (one after enrollment, and one after birth) and the infant will have one blood draw at 2-8 weeks of age. The total volume of blood required for each blood draw is 2mL from the adult participant and 1.5mL from the infant.
Fetal neuroimaging (Magnetic resonance imaging [MRI] and ultrasound) analysis | During pregnancy between 20-38 weeks gestational age
  Pregnant participants will receive one fetal MRI and ultrasound examinations during the second or third trimester. Fetal MRI will be performed on a GE 1.5 T scanner (General Electric, Milwaukee, WI) using an 8-channel head coil. Fetal ultrasound and MRI will be overseen and interpreted by fetal radiologists and neuroradiologists. Images will be evaluated for any structural abnormalities and for differences in brain maturation or size. The fronto-occipital and biparietal cerebral diameters, cerebellar vermis and diameter, and corpus callosum length will be measured. Biometric measurements and estimation of fetal cortical maturation will be compared with age-expected norms. Fetal ultrasound will be used to evaluate measurements of cerebral head circumference, biparietal diameter, body biometry, and interval growth between research scans. Fetal head circumference z-scores will be calculated from US measurements based on gestational age using the Hadlock method.
Infant neuroimaging (Magnetic resonance imaging [MRI] and ultrasound) analysis | Child age: Between 2-8 weeks
  At 2-8 weeks of age, infants will have an unsedated brain MRI and a cranial ultrasound scan. Based on investigator experience, the majority of infants can have a successful brain MRI without sedation at <6 weeks of age. The brain MRI protocol will be the standard clinical infant protocol at Children's National Hospital that includes T1, T2, susceptibility weighted imaging, and diffusion sequences. The brain MRI is without contrast.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Mulkey, MD, PhD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Participant enrollment screener — http://redcap.link/CNHLYME